CLINICAL TRIAL: NCT03422939
Title: How Dieticians Deliver Dietary Guidelines Using Portion Sizes and Time Frame
Brief Title: Dietary Guidelines, Portion Sizes, and Time Frame
Status: Completed | Type: Observational
Sponsor: Grenoble Ecole de Management (Other)
Responsible Party: Sponsor
Other Study IDs: GrenobleEM
Record Dates: First submitted 2018-01-10; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Diet Habit; Food Habits
Keywords: FBDG; dietitians; portion sizes; time frame; visual references
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Less experienced dietitians: There was no intervention, but we conducted separate analyses to identify differences according to the level of experience of the dietician. We used the median number of years of professional experience (median=8) to split the sample and create two subgroups: 1) less experienced dieticians (less than 9 years of experience; n= 225)
  Interventions: Other: there was no intervention, only separate analyses
- More experienced dietitians: and 2) more experienced dieticians (9 years of experience or more; n=215).
  Interventions: Other: there was no intervention, only separate analyses

INTERVENTIONS:
Other: there was no intervention, only separate analyses — We only conducted separate analyses to see if responses differed according to level of experience.

SUMMARY:
During the last update of the French FBDG, a survey with a representative sample of dieticians investigated 1) how to communicate portion sizes and 2) the most relevant time frame when delivering dietary guidelines. The objective was to determine how to express portion sizes and time frame for Food Based Dietary Guidelines (FBDG) using the feedback of dietitians. Data were obtained from an internet-based survey of 441 French dieticians (collected from November 24, 2013 through January 2, 2014).

DETAILED DESCRIPTION:
Background: Food Based Dietary Guidelines (FBDG) need to accessible and understandable to consumers. During the last update of the French FBDG, a survey with a representative sample of dieticians investigated 1) how to communicate portion sizes and 2) the most relevant time frame when delivering dietary guidelines.

Objective: To determine how to express portion sizes and time frame for Food Based Dietary Guidelines (FBDG) using the feedback of dietitians.

Design: Data were obtained from an internet-based survey of 441 French dieticians (collected from November 24, 2013 through January 2, 2014).

ELIGIBILITY:
Inclusion Criteria:

All members of the AFDN (French Association of Dietitians and Nutritionists) were invited to participate (n=2500 except the ones that had already participated in the pre-test n=10).

Members of the AFDN who have completed the online questionnaire were retained for analysis (n= 441).

Exclusion Criteria:

Incomplete questionnaires Participants of the pre-test (n=10)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Most participants were female (96%), were under age 45, were working in a health institution and/or had a private practice, and had, on average, 12.5 years of professional experience. Seventy-five percent received mainly adults in their practice and 62.5% received mainly patients with a health condition.
Sampling Method: Non-Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2013-11-24 (Actual); Primary Completion 2014-01-02 (Actual); Study Completion 2014-01-02 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure number of dietitians using different types of portion size and time frame | through study completion, an average of 1 month
  Open-ended questions to measure how dietitians and patients describe portion sizes and time frame

IPD SHARING:
Plan to Share IPD: Undecided